CLINICAL TRIAL: NCT02452125
Title: The Effects of Nicotine Chewing Gum on Acute Low Blood Pressure in Parkinson's Disease
Brief Title: The Effects of Nicotine Chewing Gum in Parkinson's Disease
Acronym: PD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Joanne DiFrancisco-Donoghue, Assistant Professor, New York Institute of Technology
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BHS-1118
Record Dates: First submitted 2015-05-20; First posted 2015-05-22 (Estimated); Last update posted 2017-07-28 (Actual); Status verified 2017-07

CONDITIONS: Low Blood Pressure; Parkinsons Disease
MeSH Terms: conditions — Hypotension; Parkinson Disease | interventions — Nicotine Chewing Gum

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Nicotine Gum (Experimental): Nicotine chewing gum administered for 30 minutes
  Interventions: Dietary Supplement: Nicotine gum

INTERVENTIONS:
Dietary Supplement: Nicotine gum — Nicotine chewing gum

SUMMARY:
The objective of this experiment is:

To determine if nicotine chewing gum will improve acute episodes of orthostatic hypotension in PD subjects.

DETAILED DESCRIPTION:
Subjects will be asked to sit and rest for 10 minutes. Blood pressure will be taken in this resting position after the 10 minutes.

After all inclusion criteria has been met, subjects will then wear an automated BP cuff and be administered 4mg of nicotine gum (Nicorette™). They will be instructed to use it according to manufacturer's directions and remain chewing the gum for 30 minutes. The subject will remain in a seated position and BP and HR will be recorded every 5 minutes for 30 minutes. After 30 minutes the gum will be removed and subjects will still have HR and BP monitored in the seated position for another hour every 10 minutes. All values will be compared to pretreatment values. After 120 minutes if the subject is non-symptomatic, they can go home.

ELIGIBILITY:
Inclusion Criteria:

* a diagnosis of PD
* a diastolic BP less than 90 mmHg
* and/or a systolic BP lower than 100mHg.

Exclusion Criteria:

* current tobacco users in all forms of tobacco
* severe dysphasia (difficulty swallowing)
* previous tobacco users who might be at risk for re-addiction.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2017-06-01 (Actual); Study Completion 2017-06-01 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | 90 minutes

SECONDARY OUTCOMES:
Heart Rate | 90 Minutes

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Donoghue, PhD, Principal Investigator — New York Institute of Technology
Locations (1):
- New York Institute of Technology, Old Westbury, New York, United States